CLINICAL TRIAL: NCT00371904
Title: A Prospective Open Label Randomised Multicentre Study Evaluating the Efficacy & Safety of Rituximab Given Pre-Transplant to Sensitised Renal Allograft Recipients in Addition to a "Standard" Desensitisation Regimen Consisting of PE/IVIG & MMF
Brief Title: Trial of Rituximab Given Pre-Transplant to Sensitised Live Donor Kidney Recipients
Acronym: RAPTURE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hunter and New England Health (Other)
Collaborators: Melbourne Health (Other); Princess Alexandra Hospital, Brisbane, Australia (Other); Royal Prince Alfred Hospital, Sydney, Australia (Other); Auckland City Hospital (Other Government); Monash Medical Centre (Other); Royal Perth Hospital (Other); Westmead Hospital (Unknown); Royal Adelaide Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RAPTURE
Record Dates: First submitted 2006-09-01; First posted 2006-09-04 (Estimated); Last update posted 2008-05-21 (Estimated); Status verified 2008-05

CONDITIONS: Kidney Transplantation
Keywords: Rituximab; donor; sensitised; antibody; rejection
MeSH Terms: conditions — Rejection, Psychology | interventions — Rituximab; Standard of Care

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Rituximab
- 2 (Active Comparator)
  Interventions: Drug: Standard Care

INTERVENTIONS:
Drug: Rituximab — Single dose (375 mg/m2) of rituximab to be given intravenously (IV) 14 days prior to transplantation
  Other Names: Mabthera
  Arms: 1
Drug: Standard Care — Standard care
  Arms: 2

SUMMARY:
About one third of prospective kidney transplant recipients have antibodies in their blood directed against the tissues of their only available kidney donor. Recently, "desensitisation" treatments when administered pre-transplant have allowed successful transplantation of these patients despite high rates of acute antibody mediated rejection (AAMR). The investigators propose to test in a randomised controlled trial whether rituximab, a monoclonal antibody that depletes B-lymphocytes, will safely lower antibody mediated rejection (AMR) rates when added to "standard" therapy. The investigators will also test whether rituximab enables more patients to achieve a negative crossmatch against their donor and thereby allow more transplants to proceed.

DETAILED DESCRIPTION:
This study is designed to investigate in a prospective, randomised fashion whether a single intravenous dose of rituximab (375 mg/m2) given two weeks prior to transplant, in addition to standard therapy, will allow sensitised renal transplant subjects to achieve a negative CDC crossmatch and thereby proceed to live donor transplantation. We will also evaluate whether rituximab will reduce the number of AAMR episodes in the post-transplant period, compared to controls. All eligible subjects must have a positive T- and/or B-cell CDC or flow cytometry crossmatch and have donor-specific antibodies identified by solid-phase assay at screening. All subjects will receive a standard desensitisation regimen that includes plasma exchange/IVIG + MMF before and immediately after transplantation followed by a standard care immunosuppressive regimen (IL-2R antagonist, tacrolimus, mycophenolate mofetil [MMF] and corticosteroids) after transplantation.

ELIGIBILITY:
Inclusion criteria:

1. Subjects, age > 18 years
2. Subjects receiving a single organ renal transplant from a living donor
3. Positive T-cell and/or B-cell crossmatch by complement dependent cytotoxicity (CDC) and/or positive flow cytometry crossmatch with confirmed donor-specific antibodies on solid-phase assay at screening. Positive CDC T-cell and/or B-cell crossmatch titre must be less than or equal to 1:64.
4. Subjects capable of understanding the purposes and risks of the study and who can give written informed consent

Exclusion Criteria at Study Entry (4 weeks prior to transplant):

1. Primary renal transplant lost from acute rejection less than six months prior to randomisation
2. Women of childbearing potential with a positive serum or urine pregnancy test or nursing mothers
3. Subjects with history of malignancy (other than non melanoma skin cancer that has been totally excised with no recurrence for two years)
4. Subjects with known contraindications to treatment with rituximab
5. Subjects with haemoglobin < 8.5 g/dL, WBC value of < 3000/mm3 or a platelet count of < 50,000/mm3 that is unlikely to resolve prior to randomisation
6. Subjects with a positive ABO crossmatch with donor
7. Subjects with severe diarrhoea or other gastrointestinal disorders that might interfere with the ability to absorb oral medication and is unlikely to resolve prior to randomisation
8. Subjects participating in another interventional clinical trial or requiring treatment with un-marketed investigational drugs or who would be expected to require other medications prohibited by the protocol
9. Subjects who cannot be followed for the study duration
10. Subjects with disorders or conditions that may interfere with the ability to comply with study procedures and/or requirements

Additional Exclusion Criteria at Day -2 before Transplantation:

1. All exclusion criteria as at study entry
2. Positive T- and/or B-cell CDC crossmatch at Day -2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2006-04; Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
Biopsy proven antibody mediated rejection | 12 months

SECONDARY OUTCOMES:
Elimination of donor specific antibodies (DSA) | Day - 2 , 7; Months 1, 3, 6, 9 and 12
C4d in biopsies | Day 7; Months 3 and 12
Plasma exchanges | Month 12
Death | Month 12
Treated rejection | Month 12
Graft loss | Months 3, 6 and 12
Treatment failure | Months 6 and 12
Calculation of glomerular filtration rate (GFR) | Months 1 - 12
Slope of 1/serum creatinine (Ser. Cr) | Months 6 and 12
24-hour U protein | Months 3 and 12
Safety | Month 12
Cancer and infections | Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Paul R Trevillian, MBBS, FRACP, Study Chair — Newcastle Transplant Unit, John Hunter Hospital; Solomon Cohney, MBBS, FRACP, PhD, Study Chair — Melbourne Health
Locations (3):
- Australia (3):
  - Newcastle Transplant Unit, John Hunter Hospital, Newcastle, New South Wales
  - Monash Medical Centre, Clayton, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria